CLINICAL TRIAL: NCT04892121
Title: The Efficiency of a Warm-up Prevention Program in Volleyball Players
Brief Title: Prevention in Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Camille Tooth, Principal Investigator, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Prevention VB
Record Dates: First submitted 2020-03-09; First posted 2021-05-19 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Prevention
Keywords: prevention, shoulder, exercises, volleyball
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The teams in the intervention group will have to follow a warm-up prevention program twice a week
  Interventions: Other: Prevention exercises
- Control group (No Intervention): The teams in the control group will have to reply each month to a questionnaire about the potential injuries they experienced during the previous month.

INTERVENTIONS:
Other: Prevention exercises — Participants will have to follow a warm-up prevention program (15 minutes) twice a week
  Arms: Intervention group

SUMMARY:
The objective of this study is to assess the interest and the efficiency of a warm-up prevention program on the prevalence of shoulder injuries in amateur volleyball players.

Around ten teams will be included in the study. They will be divided into two groups (blind): an intervention group and a control group.

A warm-up prevention program will implemented in the teams of intervention group. This program will have to be followed twice a week, at the beginning of the training session.

In both groups, shoulder injuries will be registered each month by an online questionnaire.

DETAILED DESCRIPTION:
Around ten teams will be recruted among the clubs in the Province of Liege. They will be divided into two groups (blind): an intervention group and a control group.

Each month, both groups will be asked to fill in a form with the potential injuries they experienced during the past month.

* Intervention group :

All the teams included in the intervention group will be asked to follow a warm-up prevention program (about 15 minutes) at least twice a week, at the beginning of the training session.

At the beginning of the season, one experimenter will go to the different clubs in order to present the program, to explain the exercises and to correct the players while doint the exercises.

During the season, the same experimenter will go to the clubs at regular intervals to make sure that the players are well doing the program and to assess the compliance.

- Control group :

The objective of the control group is to estimate the prevalence of shoulder injuries in a group without any prevention implementation. The players of this group will jus have to answer the monthly questionnaire about the potential injuries they experienced during the previous month.

ELIGIBILITY:
Inclusion Criteria:

* volleyball players in Provincial level (P1-P2)
* practicing volleyball at least 4 hours in a week
* no "prevention routines"

Exclusion Criteria:

* having a prevention program

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 93 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of shoulder injuries | through study completion, an average of 1 year
  The number of injuries the players experienced during the season
Compliance with the program | through study completion, an average of 1 year
  The number of time the players did the program during each month

CONTACTS AND LOCATIONS:
Locations (1):
- Fédération de Volleyball Wallonie-Bruxelles, Namur, Belgium

IPD SHARING:
Plan to Share IPD: No